CLINICAL TRIAL: NCT04064645
Title: BiOSENCY Bora Band Respiration Rate Development and Validation Study
Brief Title: Bora Band Respiration Rate Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosency (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR2019-319
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Respiratory rate accuracy measurement (Experimental)
  Interventions: Device: Measurement of respiratory rate with DUT and comparison with reference

INTERVENTIONS:
Device: Measurement of respiratory rate with DUT and comparison with reference — The subject will follow the paced breathing app, once a stable Respiration Rate at the natural rate (without the breathing app) is captured. The breathing pattern on the app will be set to begin near the normal Respiration Rate of the subject and continue to go down by five intervals until reaching the Respiration Rate of 5 bpm. After that, we will pick back up at the rate above the subject's normal Respiration Rate and continue upwards until reaching 50 bpm or as high as the subject can tolerate up to 50 bpm.
  The respiratory rate will be monitored simultaneously with an EtCo2 (Reference) and the BORA BAND™ wristband monitoring system, Device Under Test. These data will be continuously recorded electronically. Additional study notes that describe conditions of the test as well as deviations, device issues and any adverse events will be recorded in written documentation.

SUMMARY:
The purpose of this study is to conduct a Respiratory Rate accuracy validation comparing the BORA BAND™ Wristband Monitoring System to the Reference. Respiratory Rate will be compared to an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda). The testing will be conducted in two phases. The first phase will be an initial data collection to assist in the algorithm development of respiration rate. Upon a successful Phase one performance, the second phase will be the Respiratory Rate Validation conducted at a different period in time.

DETAILED DESCRIPTION:
For phase 1, there will be 5 to 6 volunteer test subjects. For the final validation phase, there will be a minimum of 20 volunteer test subjects. All subjects will be 18 or older and selected to represent a range of body types including small, average, muscular, and large with a range of BMI's.

Each subject will be connected to a commonly used, FDA cleared ECG Impedance monitor (to be used for informational purposes) and an End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) and BiOSENCY BORA BAND™ wristband monitoring system. The end tidal CO2 monitor will be attached to the patient to determine performance of respiratory rate metrics (Reference). Each subject will be instrumented with a mouthpiece that allows for measurement of the end tidal carbon dioxide (EtCO2) respiratory rate (Reference) and tidal volume.

A range of stable respiratory rates will be elicited from each volunteer test subject. The rates will be approximately 5, 10, 15, 20, 25, 30, 35, 40, 45 and 50 breaths per minute; with some natural variation from these exact numbers. Paced breathing app will be used. Not all subjects will be able to breathe at a constant level for every rate.

The respiratory rate will be measured simultaneously with EtCO2 (Reference) and the Devices Under Test.

For the data analysis, the EtCO2 monitor will be used to assess the stability of the data. If the respiratory rate varies by more than +3 bpm during a one-minute period of the target respiration rates, then the data for that period will be considered unstable and removed from analysis.

To 'Pass' this test the BiOSENCY BORA BAND™ wristband (Device Under Test) must demonstrate a Respiratory Rate of ≤3 when compared to the Reference End tidal carbon dioxide monitor.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is adult over 18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker
* Male or female of any race
* Wrist circumference with the range of 5.5-8 inches (13 to 21cm)

Exclusion Criteria:

* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoo in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
* Cancer / chemotherapy
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of BORA Band respiratory rate measurements versus reference end-tidal CO2 | 5 days
  Accuracy of the BORA Band respiratory rate measurement as compared to reference end-tidal CO2.
  Results shall include:
  * Respiratory rate root mean square accuracy of BORA Band
  * Respiratory rate bias of BORA Band

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark Laboratory, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No